CLINICAL TRIAL: NCT04903288
Title: An Open-Label Trial to Address the Safety of the SmartFlow MR-Compatible Ventricular Cannula for Administering Eladocagene Exuparvovec to Pediatric Subjects
Brief Title: A Study of SmartFlow Magnetic Resonance (MR) Compatible Ventricular Cannula for Administering Eladocagene Exuparvovec to Pediatric Participants
Status: Active, not recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: PTC Therapeutics (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: PTC-AADC-GT-002
Record Dates: First submitted 2021-05-21; First posted 2021-05-26 (Actual); Results first posted 2025-01-01 (Actual); Last update posted 2026-01-30 (Actual); Status verified 2026-01

CONDITIONS: AADC Deficiency
Keywords: AADC Deficiency gene therapy
MeSH Terms: conditions — Aromatic amino acid decarboxylase deficiency

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: Yes

ARMS (1):
- Eladocagene Exuparvovec (Experimental): Participants will receive eladocagene exuparvovec intraoperatively at 1.8×10^11 vector genomes (vg) via SmartFlow® MR Compatible Ventricular Cannula in a single operative session. Participants will receive standard of care for their AADC deficiency during the study.
  Interventions: Genetic: Eladocagene Exuparvovec

INTERVENTIONS:
Genetic: Eladocagene Exuparvovec — Four 0.08 milliliters (mL) infusions at a dose of 0.45×10^11 vg and a volume of 80 microliters (μl) per site to 4 sites (2 per putamen), for the total dose of 1.8×10^11 vg and a total volume of 320 μl per participant.
  Other Names: KEBILIDI™

SUMMARY:
This study will have a trial phase, extension phase, and a long-term extension phase. The primary objectives of the trial phase are to assess the pharmacodynamics (PD) of eladocagene exuparvovec treatment by evaluation of homovanillic acid (HVA) levels and to assess the safety of the SmartFlow® magnetic resonance (MR) Compatible Ventricular Cannula for administering eladocagene exuparvovec to pediatric participants with aromatic L-amino acid decarboxylase (AADC) deficiency. The extension phase is designed to capture additional clinical information for eladocagene exuparvovec through study evaluations, changes in motor development, AADC-specific symptoms, and other PD measures. The long-term extension phase is designed to capture long-term safety and efficacy data from participants treated with eladocagene exuparvovec.

ELIGIBILITY:
Inclusion Criteria:

* Pediatric participants must have genetically-confirmed AADC deficiency with typical clinical characteristics and decreased AADC enzyme activity in plasma.
* Cranium sufficiently developed to allow placement of ClearPoint® system for stereotactic surgery.
* Persistent neurological defects secondary to AADC deficiency despite standard medical therapy (dopamine agonists, monoamine oxidase inhibitor, pyridoxine, or other forms of vitamin B6) in the opinion of the investigator.
* Unable to ambulate independently (with or without assistive device).
* Baseline hematology, chemistry, and coagulation values within the normal pediatric laboratory value ranges, unless in the investigator's opinion the out of range values are not clinically significant with respect to the participant's suitability for surgery.
* Participant must test negative for coronavirus disease of 2019 (COVID-19) a maximum of 72 hours prior to receiving gene therapy.
* Participant must be on stable dosage for 3 months prior to baseline for all medications related to treatment of AADC deficiency, including dopamine agonists, monoamine oxidase inhibitors, anticholinergic drugs, and vitamin B6.
* Females of childbearing potential must have a negative pregnancy test at screening and baseline and agree to abstinence or double-barrier form of contraception for the duration of the study following discharge from the hospital (acceptable methods will be determined by the site).
* Males sexually active with females of childbearing potential must agree to use a barrier method of birth control during the study following discharge from the hospital.
* Parent(s)/legal guardian(s) of the participant must agree to comply with the requirements of the study, including the need for frequent and prolonged follow up.
* Parent(s)/legal guardian(s) with custody of the participant must give their consent for the participant to enroll in the study.

Exclusion Criteria:

* The participant has presence of other significant medical or neurological conditions that would create an unacceptable operative or anesthetic risk.
* Participants with pyridoxine 5'-phosphate oxidase or tetrahydrobiopterin (BH4) deficiency.
* Contraindication for imaging studies (computed tomography [CT] scan, PET or magnetic resonance imaging [MRI]), including sedation limitations or metal that would interfere with a brain MRI.
* Anti-adeno-associated virus, serotype 2 (anti-AAV2) antibody titer higher than 1:1200 or >1 optical density value by enzyme-linked immunosorbent assay.
* Participants who have received treatment with other experimental therapies within the last 24 weeks prior to planned gene therapy administration, or any treatment ever with a gene therapy.
* Evidence of a clinically active infection.
* Females who are pregnant or breast feeding.

Ages: 1 Year to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 13 (Actual)
Dates: Start 2021-05-12 (Actual); Primary Completion 2023-05-22 (Actual); Study Completion 2028-04-30 (Estimated)

CONTACTS AND LOCATIONS:
Locations (6):
- United States (4):
  - Boston Children's Hospital, Boston, Massachusetts
  - Duke University Hospital, Durham, North Carolina
  - Cincinnati Children's Hospital Medical Center, Cincinnati, Ohio
  - Texas Children's Hospital, Houston, Texas
- Chaim Sheba Medical Center, Ramat Gan, Israel
- National Taiwan University Hospital, Department of Pediatrics and Medical Genetics, Taipei, Taiwan

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: The study is ongoing. Only primary analysis results are reported. Final results will be reported after completion of study.
Groups:
- Eladocagene Exuparvovec: Participants received eladocagene exuparvovec intraoperatively at 1.8×10^11 vector genomes (vg) via SmartFlow® MR Compatible Ventricular Cannula in a single operative session. Participants received standard of care for their aromatic L-amino acid decarboxylase (AADC) deficiency during the study.
Period: Trial Phase (8 Weeks)
Arm/Group | Eladocagene Exuparvovec
Started | 13
Received at Least 1 Dose of Study Drug | 13
Completed | 13
Not Completed | 0
Period: Extension Phase (48 Weeks)
Arm/Group | Eladocagene Exuparvovec
Started | 13
Completed | 9
Not Completed | 4
Not completed — Withdrawal by Subject | 1
Not completed — Ongoing in the Study | 3
Period: Long-Term Extension Phase (60 Months)
Arm/Group | Eladocagene Exuparvovec
Started | 7
Completed | 0
Not Completed | 7
Not completed — Withdrawal by Subject | 1
Not completed — Ongoing in the Study | 6

BASELINE CHARACTERISTICS:
Population: The safety population included all participants enrolled in the study who have received any amount of study drug.
Groups:
- Eladocagene Exuparvovec: Participants received eladocagene exuparvovec intraoperatively at 1.8×10^11 vg via SmartFlow® MR Compatible Ventricular Cannula in a single operative session. Participants received standard of care for their AADC deficiency during the study.
Arm/Group | Eladocagene Exuparvovec
Number analyzed (Participants) | 13
Age, Continuous [Mean (Standard Deviation); unit: months] | 45.2 (29.48)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 7
  Male | 6
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 2
  Not Hispanic or Latino | 10
  Unknown or Not Reported | 1
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 10
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 2
  More than one race | 0
  Unknown or Not Reported | 1
Homovanillic Acid (HVA) Metabolite Level [Mean (Standard Deviation); unit: nanomoles (nmol)/liter (L)] — HVA is a main metabolite of dopamine and HVA cerebrospinal fluid (CSF) levels are recognized as a proxy for dopamine levels in the brain.
  nanomoles (nmol)/liter (L) | 22.54 (32.34)

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline in HVA Metabolite Level at the End of the Trial Phase
Description: HVA is a main metabolite of dopamine and HVA CSF levels are recognized as a proxy for dopamine levels in the brain.
Time Frame: Baseline (Day 1), Week 8
Population: The safety population included all participants enrolled in the study who have received any amount of study drug. 'Overall number of participants analyzed' = participants evaluable for this outcome measure.
Measure: Mean (Standard Deviation); unit: nmol/L
Arm/Group | Eladocagene Exuparvovec
Number analyzed (Participants) | 12
nmol/L | 29.53 (12.93)

2. Primary Outcome: Number of Participants With Adverse Events (AEs) Associated With the Surgical Administration of Eladocagene Exuparvovec Using the SmartFlow® MR-Compatible Ventricular Cannula
Description: An AE is any untoward medical occurrence associated with the use of a drug in humans, whether or not it is considered related to the drug. An AE can therefore be any unfavorable and unintended sign (including an abnormal laboratory finding), symptom, or disease in a study participant who was administered gene therapy in this study. Number of participants with AEs related to the SmartFlow MR-compatible ventricular cannula used to administer eladocagene exuparvovec to pediatric participants at the end of Trial Phase (8 weeks after administration) are reported. A summary of serious and all other non-serious adverse events regardless of causality is located in the Reported Adverse Events module."
Time Frame: Baseline (Day 1) up to Week 8
Population: The safety population included all participants enrolled in the study who have received any amount of study drug.
Measure: Count of Participants; unit: Participants
Arm/Group | Eladocagene Exuparvovec
Number analyzed (Participants) | 13
Participants | 0

3. Secondary Outcome: Change From Baseline in Neurotransmitter Cerebrospinal Fluid (CSF) Metabolite HVA at Week 48
Time Frame: Baseline (Day 1), Week 48
Reporting Status: Not Posted, anticipated posting 2029-04

4. Secondary Outcome: Change From Baseline in Positron Emission Tomography (PET) Imaging of Putaminal-Specific L-6-[18F] Fluoro-3,4-Dihydroxyphenylalnine (18F-DOPA) PET Uptake at the End of the Trial Phase (Week 8) and the Extension Phase (Week 48)
Time Frame: Baseline (Day 1), Week 8, Week 48
Reporting Status: Not Posted, anticipated posting 2029-04

5. Secondary Outcome: Change From Baseline in Neurotransmitter CSF Metabolites 5-hydroxyindoleacetic Acid (5-HIAA), and 3-O-methyldopa (3-OMD) at Weeks 8 and 48
Time Frame: Baseline (Day 1), Weeks 8 and 48
Reporting Status: Not Posted, anticipated posting 2029-04

6. Secondary Outcome: Number of Participants Who Attain Motor Milestones
Time Frame: Baseline (Day 1) up to Week 260
Reporting Status: Not Posted, anticipated posting 2029-04

7. Secondary Outcome: Change in Peabody Developmental Motor Scale, Second Edition (PDMS-2)
Time Frame: Baseline (Day 1), Week 260
Reporting Status: Not Posted, anticipated posting 2029-04

8. Secondary Outcome: Change in Bayley Scale of Infant Development, Third Edition (Bayley-III)
Time Frame: Baseline (Day 1), Week 260
Reporting Status: Not Posted, anticipated posting 2029-04

9. Secondary Outcome: Change in EuroQol-5 Dimensions Youth Version (EQ-5D-Y)
Time Frame: Baseline (Day 1), Week 260
Reporting Status: Not Posted, anticipated posting 2029-04

10. Secondary Outcome: Change in Body Weight
Time Frame: Baseline (Day 1), Week 260
Reporting Status: Not Posted, anticipated posting 2029-04

11. Secondary Outcome: Number of Participants With AADC-Specific Symptoms
Time Frame: Baseline (Day 1) up to Week 260
Reporting Status: Not Posted, anticipated posting 2029-04

12. Secondary Outcome: "Number of Participants With Treatment-Emergent Adverse Events (TEAEs) "
Time Frame: Baseline (Day 1) up to Week 260
Reporting Status: Not Posted, anticipated posting 2029-04

ADVERSE EVENTS:
Time Frame: Baseline (Day 1) up to the interim data cut-off date (up to 897 days)
Description: The safety population included all participants enrolled in the study who have received any amount of study drug.
Arm/Group | Eladocagene Exuparvovec
All-Cause Mortality (participants affected / at risk) | 0/13
Serious Adverse Events (participants affected / at risk) | 9/13
Other Adverse Events (participants affected / at risk) | 13/13
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Eladocagene Exuparvovec (N=13)
Bradycardia (Cardiac disorders) | 1
Vomiting (Gastrointestinal disorders) | 1
Pyrexia (General disorders) | 1
Bacterial infection (Infections and infestations) | 1
COVID-19 (Infections and infestations) | 1
Metapneumovirus pneumonia (Infections and infestations) | 1
Pneumonia (Infections and infestations) | 3
Pneumonia viral (Infections and infestations) | 1
Urinary tract infection (Infections and infestations) | 1
Dyskinesia (Nervous system disorders) | 1
Seizure (Nervous system disorders) | 1
Bronchospasm (Respiratory, thoracic and mediastinal disorders) | 1
Respiratory arrest (Respiratory, thoracic and mediastinal disorders) | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Eladocagene Exuparvovec (N=13)
Anaemia (Blood and lymphatic system disorders) | 4
Lymphadenopathy (Blood and lymphatic system disorders) | 1
Tachycardia (Cardiac disorders) | 1
Dry eye (Eye disorders) | 1
Eye swelling (Eye disorders) | 2
Ocular hyperaemia (Eye disorders) | 1
Oculogyric crisis (Eye disorders) | 2
Periorbital oedema (Eye disorders) | 1
Anal fissure (Gastrointestinal disorders) | 1
Constipation (Gastrointestinal disorders) | 1
Diarrhoea (Gastrointestinal disorders) | 8
Discoloured vomit (Gastrointestinal disorders) | 1
Dysphagia (Gastrointestinal disorders) | 1
Flatulence (Gastrointestinal disorders) | 1
Gastrointestinal haemorrhage (Gastrointestinal disorders) | 1
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 1
Haematemesis (Gastrointestinal disorders) | 1
Salivary hypersecretion (Gastrointestinal disorders) | 3
Stomatitis (Gastrointestinal disorders) | 1
Upper gastrointestinal haemorrhage (Gastrointestinal disorders) | 1
Vomiting (Gastrointestinal disorders) | 4
Face oedema (General disorders) | 1
Infusion site bruising (General disorders) | 1
Injury associated with device (General disorders) | 1
Puncture site pain (General disorders) | 1
Pyrexia (General disorders) | 10
COVID-19 (Infections and infestations) | 2
Clostridium difficile infection (Infections and infestations) | 1
Conjunctivitis bacterial (Infections and infestations) | 1
Ear infection (Infections and infestations) | 1
Gastroenteritis viral (Infections and infestations) | 1
Impetigo (Infections and infestations) | 1
Influenza (Infections and infestations) | 3
Nasopharyngitis (Infections and infestations) | 4
Otitis media (Infections and infestations) | 1
Otitis media acute (Infections and infestations) | 1
Pneumonia (Infections and infestations) | 2
Pneumonia aspiration (Infections and infestations) | 1
Post viral fatigue syndrome (Infections and infestations) | 1
Rhinovirus infection (Infections and infestations) | 1
Tinea cruris (Infections and infestations) | 1
Upper respiratory tract infection (Infections and infestations) | 3
Viral upper respiratory tract infection (Infections and infestations) | 1
Contusion (Injury, poisoning and procedural complications) | 2
Fall (Injury, poisoning and procedural complications) | 1
Forearm fracture (Injury, poisoning and procedural complications) | 1
Incision site haemorrhage (Injury, poisoning and procedural complications) | 1
Post procedural hypotension (Injury, poisoning and procedural complications) | 1
Scratch (Injury, poisoning and procedural complications) | 2
Skin abrasion (Injury, poisoning and procedural complications) | 1
Skin pressure mark (Injury, poisoning and procedural complications) | 1
Stoma site discharge (Injury, poisoning and procedural complications) | 1
Alanine aminotransferase increased (Investigations) | 1
Aspartate aminotransferase increased (Investigations) | 1
Blood alkaline phosphatase increased (Investigations) | 1
Blood bicarbonate decreased (Investigations) | 1
Blood creatinine decreased (Investigations) | 1
Blood potassium decreased (Investigations) | 1
Eosinophil count increased (Investigations) | 1
Heart rate increased (Investigations) | 1
Lymphocyte count increased (Investigations) | 1
SARS-CoV-2 test positive (Investigations) | 2
Viral test positive (Investigations) | 2
White blood cell count increased (Investigations) | 1
Decreased appetite (Metabolism and nutrition disorders) | 1
Hyperglycaemia (Metabolism and nutrition disorders) | 1
Hypocalcaemia (Metabolism and nutrition disorders) | 1
Hypoglycaemia (Metabolism and nutrition disorders) | 2
Hypokalaemia (Metabolism and nutrition disorders) | 3
Hypomagnesaemia (Metabolism and nutrition disorders) | 2
Hypophosphataemia (Metabolism and nutrition disorders) | 3
Polydipsia (Metabolism and nutrition disorders) | 1
Dyskinesia (Nervous system disorders) | 10
Myoclonus (Nervous system disorders) | 1
Insomnia (Psychiatric disorders) | 3
Atelectasis (Respiratory, thoracic and mediastinal disorders) | 1
Cough (Respiratory, thoracic and mediastinal disorders) | 5
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 1
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 1
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 2
Increased upper airway secretion (Respiratory, thoracic and mediastinal disorders) | 1
Lung hyperinflation (Respiratory, thoracic and mediastinal disorders) | 1
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 3
Rhinitis allergic (Respiratory, thoracic and mediastinal disorders) | 1
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 3
Sinus congestion (Respiratory, thoracic and mediastinal disorders) | 1
Tachypnoea (Respiratory, thoracic and mediastinal disorders) | 1
Upper respiratory tract congestion (Respiratory, thoracic and mediastinal disorders) | 1
Dermatitis atopic (Skin and subcutaneous tissue disorders) | 1
Dermatitis diaper (Skin and subcutaneous tissue disorders) | 5
Eczema (Skin and subcutaneous tissue disorders) | 1
Rash (Skin and subcutaneous tissue disorders) | 1
Skin lesion inflammation (Skin and subcutaneous tissue disorders) | 1
Cyanosis (Vascular disorders) | 1
Hypotension (Vascular disorders) | 4

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The Sponsor can review results and/or communications prior to public release and can embargo communications regarding trial results for a period that is up to 180 days from the time submitted to the sponsor for review. The sponsor may consult with the PI to require changes to the communication or extend the embargo.

DOCUMENTS (2):
  • Study Protocol (2023-09-01): https://cdn.clinicaltrials.gov/large-docs/88/NCT04903288/Prot_000.pdf
  • Statistical Analysis Plan (2024-01-24): https://cdn.clinicaltrials.gov/large-docs/88/NCT04903288/SAP_001.pdf